CLINICAL TRIAL: NCT06314672
Title: The Ohio State University Connecting Underrepresented Populations to Clinical Trials (CUSP2CT) Project
Brief Title: Outreach Project to Connect Underrepresented Populations to Clinical Trials at Ohio State University, CUSP2CT Project Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-22318; NCI-2023-02217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA274999 (NIH)
Record Dates: First submitted 2023-10-31; First posted 2024-03-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (interview, discussion, review, AEP, education) (Experimental): Community members, clinic staff, and providers undergo in-depth interview for intervention development on study. Researchers review baseline data on referral patterns and accrual of racial and ethnic minorities to clinical trials in each clinic site. Providers, clinical staff, and research team participate in implementation discussion. AEP strategies developed and initiated in one OSUCCC/James clinic. Providers and community members participate in educational sessions on study. (Year 1)
  Interventions: Procedure: Accrual; Procedure: Discussion; Other: Educational Activity; Other: Interview; Other: Review; Other: Survey Administration
- Phase II (AEP, education, interviews) (Experimental): Participants participate in the AEP in the remaining clinics at OSUCCC/James and community clinics on study. Community members and providers participate in culturally tailored educational activities. Providers, patients, and community members participate in interviews to explore current barriers to referral and participation on study. (Years 2-4)
  Interventions: Procedure: Accrual; Other: Educational Activity; Other: Interview; Other: Survey Administration
- Phase III (interview) (Experimental): Providers, clinic staff, patients, and community members participate in interviews to explore current barriers to referral and participation. (Year 5)
  Interventions: Other: Interview

INTERVENTIONS:
Procedure: Accrual — Participate in AEP
  Arms: Phase I (interview, discussion, review, AEP, education); Phase II (AEP, education, interviews)
Procedure: Discussion — Participate in implementation discussions
  Other Names: Discuss
  Arms: Phase I (interview, discussion, review, AEP, education)
Other: Educational Activity — Participate in educational sessions/activities
  Arms: Phase I (interview, discussion, review, AEP, education); Phase II (AEP, education, interviews)
Other: Interview — Undergo interview
Other: Review — Undergo data capture review
  Arms: Phase I (interview, discussion, review, AEP, education)
Other: Survey Administration — Ancillary studies
  Arms: Phase I (interview, discussion, review, AEP, education); Phase II (AEP, education, interviews)

SUMMARY:
This clinical trial tests the impact of the The Ohio State University Connecting Underrepresented Populations to Clinical Trials (CUSP2CT) project on clinical trial referrals and enrollment in racial/ethnic minorities. Progress in cancer prevention, detection and treatment can only be made by identifying and validating new and improved methods, compounds and modalities in clinical trials. Unfortunately, participation in clinical trials is not equal across all racial and ethnic groups, limiting progress against cancer in all population groups and further widening the disparity gap. To change this picture, concerted effort needs to be directed both at the communities at risk for being left out of trials and the systems that cause the disparities at all levels involved in accrual to clinical trials. The CUSP2CT project may have the potential to increase referral and accrual of racial/ethnic minorities to prevention/control and treatment trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a baseline assessment of referral patterns and accrual of racial and ethnic minorities to clinical trials at Ohio State University Comprehensive Cancer Center (OSUCCC) by cancer disease group (breast, gastrointestinal, genitourinary, thoracic, hematologic,and others) and examine factors at the system (i.e., eligible clinical trial protocol, clinic context and culture), provider (trial discussed with patient) and patient levels (agreed or refused participation) that influence referral and accrual. (Phase I) II. Implement a multi-level intervention in a stepped wedge design in referral in 10 counties in the OSUCCC catchment area using the Accrual to Clinical Trials framework. (Phase II) III. Evaluate the impact of the intervention on referral (primary outcome) and accrual (secondary outcomes) to clinical trials. (Phase III)

OUTLINE: Counties are cluster randomized to 1 of 3 steps in Phase II of the study.

PHASE I (DEVELOPMENT): Community members, clinic staff, and providers undergo in-depth interview for intervention development on study. Researchers review baseline data on referral patterns and accrual of racial and ethnic minorities to clinical trials in each clinic site. Providers, clinical staff, and research team participate in implementation discussion. Accrual enhancement program (AEP) strategies developed and initiated in one OSUCCC/James clinic. Providers and community members participate in educational sessions on study. (Year 1)

PHASE II (IMPLEMENTATION): Participants participate in the AEP in the remaining clinics at OSUCCC/James and community clinics on study. Community members and providers participate in culturally tailored educational activities. Providers, patients, and community members participate in interviews to explore current barriers to referral and participation on study. (Years 2-4)

PHASE III (EVALUATION): Providers, clinic staff, patients, and community members participate in interviews to explore current barriers to referral and participation. (Year 5)

ELIGIBILITY:
Inclusion Criteria:

* Phase I: 9 counties in the OSUCCC catchment area
* Phase II: Patients, providers, and hospital systems/referral centers that directly addresses challenges identified in Phase I
* Phase II: The project will involve the OSUCCC, the OSU James Cancer Network sites and the Columbus and Dayton NCORP sites

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in referral rate to clinical trials (CTs) (short-term outcomes) | Baseline to 24 months
  Calculate change in clinical trial referrals
Change in accrual of minorities to CTs (short-term outcomes) | Baseline to 24 months
  Calculate the change in clinical trial minority enrollments
CT accrual and retention due to patient navigation (short-term outcomes) | Baseline to 24 months
  Calculate accrual and retention rates
Identification of program gaps in trial accrual (long-term outcomes) | Up to 24 months
  Define gaps in trial accrual
Uptake of program in other clinics (long-germ outcomes) | Up to 24 months
  Calculate the number of clinics who adapt program

SECONDARY OUTCOMES:
Probability of trial enrollment and retention | Up to 24 months
  Recent regression models used for stepped wedge designs that flexibly model the effect curve of the intervention over time. Effect estimates and 95% confidence intervals will accompany significance tests, and graphical displays of the final effect curve will aid in understanding the efficacy of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu